CLINICAL TRIAL: NCT04084379
Title: Implementation Strategy of Bio-molecular Techniques for Early Diagnose of Congenital Syphilis and Chagas Diseases in Context of ETMIplus Program, OPS/OMS. Multicentric Study
Brief Title: Implementation Strategy of Bio-molecular Techniques for Early Diagnose of Congenital Syphilis and Chagas Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Dr Jaime Altcheh, Principal Investigator, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: ETMIplus ChC/SiC
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Chagas Disease; Syphilis
Keywords: congenital chagas disease; congenital syphilis; Chagas PCR diagnose; Syphilis PCR diagnose; Children
MeSH Terms: conditions — Chagas Disease; Syphilis; Syphilis, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chagas disease and syphilis are considered a mayor public health problem worldwide. Both pathologies affect socio-economic vulnerable population and they are both transmitted congenitally, causing an alarming increasing number of infected newborns. The current diagnostic methods for these diseases are based on serology follow-up until 8 to 10 months from birth, which considering the population usually involved and their scarce resources, usually translates in loosing continuity in their controls and follow-up.

Chagas prevalence in pregnant women is 4% with an incidence of Congenital Chagas disease of 1500 annual cases. From those, only 1 third are diagnosed. In the investigators and other authors experience, the detection of DNA of Trypanosoma cruzi by PCR shows an elevation of parasitemia at birth, with a peak at the first month of life.

Syphilis is a re-emergent pathology, preventable and curable when diagnose is achieved early at the beginning of pregnancy.. The cost-effectiveness of performing screening for this infection is widely demonstrated, preventing high morbi-mortality for children when applied to pregnant women.

For both syphilis and Chagas diagnosis, there are some studies comparing PCR follow-up with conventional serology, but none were validated and there is still need to bring more evidence in order to modify current practice. The investigators propose a sequential study of PCR for Tryipanosoma cruzi and Treponema pallidum from birth, believing this will increase sensitivity of congenital Chagas and syphilis diagnose and improve follow-up of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Child under 1 year of age, born from mother positive for syphilis not treated or inadequately treated during pregnancy
* Patients with acquired syphilis
* Child under 1 year of age, born from mother with positive serology test for Chagas

Exclusion Criteria:

* Patients who had received treatment for syphilis or Chagas previously
* Patients who are not able to complete scheduled visits
* Other diseases that could difficult implementation of this protocol or results interpretation.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Population of this study are children born from mother positive for syphilis or Chagas diseases, with congenital infection suspected and children with acquired syphilis.
  They will be recruited at five centers from different geographical areas of Argentina
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Implementation of Bio-molecular Techniques (PCR) for Early Diagnose of Congenital Syphilis and Chagas Diseases | 2 years
  Evaluate PCR sensitivity, specificity, PPV and NPP in diagnose of congenital syphilis and congenital Chagas diseases and compare it with current methods. The investigators will measure PCR titles during one year in each patient, and then compare results with serologies, in order to assess if PCR positivization and negativization occurs earlier than current methods. This may allow physicians to shorten time required for follow-up in these patients.

SECONDARY OUTCOMES:
Implementation of Bio-molecular Techniques (PCR) as terapeutic response biomarker for Congenital Syphilis and Chagas Disease | 2 years
  Investigators will evaluate the utility of PCR as an early biomarker of terapeutic response and compare it to serology for T.pallidum and T. cruzi during and after treatment. This could prevent unnecessary prolonged treatments, and could also allow early diagnose for treatment failures.
Identification of different genotypes of T.pallidum in samples to create a database of T.pallidum genotypes | 2 years
  Identification of different genotypes of T.pallidum in samples taken from active skin lessions and blood samples, in order to create a data base of T.pallidum genotypes causing congenital syphilis and acquired syphilis

CONTACTS AND LOCATIONS:
Locations (1):
- Parasitology Division, Children's Hospital "R Gutierrez" of Buenos Aires, Buenos Aires, Argentina